CLINICAL TRIAL: NCT02214836
Title: Ultrasound Imaging of Kidney Stones and Lithotripsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Bailey, Research Engineer, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00003444; P01DK043881 (NIH); CDMRP-SC220095 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2014-08-07; First posted 2014-08-12 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Kidney Stones; Nephrolithiasis; Urolithiasis; Ureter Stones
Keywords: kidney stones; ultrasound imaging; ureter stones
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis; Urolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Kidney stones (Experimental): Device: Verasonics Data Acquisition System (VDAS)
  Other Names:
  Verasonics Data Acquisition System (VDAS) Verasonics Ultrasound Engine Subjects will be imaged the Verasonics Data Acquisition System (VDAS) using conventional clinical outputs within FDA limits. The image processing has been modified.
  Subjects in this arm will be imaged by ultrasound by the VDAS. Stone location and size will be determined and compared to clinical determination of stone location and size.
  Interventions: Device: Verasonics Data Acquisition System (VDAS)

INTERVENTIONS:
Device: Verasonics Data Acquisition System (VDAS) — Subjects will be imaged the Verasonics Data Acquisition System (VDAS) using conventional clinical outputs within FDA limits. The image processing has been modified. Stone location and size will be determined and compared to clinical determination of stone location and size.
  Other Names: Verasonics Ultrasound Engine

SUMMARY:
The purpose of this study is to determine whether new software processing of ultrasound images can improve detection and size determination of kidney stones.

DETAILED DESCRIPTION:
The purpose of our research is to improve the ability to see kidney stones with ultrasound imaging. Specifically, we are testing how well new stone specific processing can find stones and show their size. Ultimately, better imaging can improve the care of future patients.

Patients with kidney stones or undergoing surgery for kidney stones will be recruited and consented.

We will image the kidney and ureter stones of consented subjects. We will place a water-based gel and ultrasound probe against the subject's skin on the back, sides, and abdomen. We will save the images and the raw electrical signals received from the probe and used to make the images. The images will be used to estimate the location and size of kidney stones in the kidney or ureter. The size and location will also be determined from x-ray and ultrasound images and reports already in the subject's medical record. And for recruited subjects who are already undergoing surgery in an existing clinical not research procedure, the surgeon will also measure location and size of stones seen in surgery. All these measurements of size and location of kidney stones will be compared to test the accuracy of the new ultrasound image processing.

After the examination, we will not ask anything more of subjects, but we will collect some information from their existing medical records. This information includes existing images of your stones, size of stones, location of stones, number of stones, type of stones, and treatment records. We will also record your weight, height, race, and ethnicity. Not all this information may be available. We will use what information is available. This additional information is used to test how well our ultrasound exam did. It also shows if we do better with certain groups of patients, for example, for certain stone types or body sizes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with kidney stones that are visible on x-ray (i.e., calcium stones)
* Current CT scan within the 90-day pre-operative period
* Able to give informed consent
* Age 21 years or older

Exclusion Criteria:

* Inability to give informed consent
* Age less than 21 years
* Stones not visible on x-ray
* Patients with systemic disease or renal anatomical disorders (RTA, primary hyperparathyroidism, sarcoidosis, enteric hyperoxaluria, medullary sponge kidney)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number and location of stones identified on research ultrasound vs. clinically. The outcome measured will be the accuracy new ultrasound images versus existing clinical data. | Research data are collected on Day 1 (the day of the research imaging procedure). Clinical data are also available on Day 1. Clinical data will be downloaded by Day 7, and comparison will be made by Day 14.
  Number and location of stones will be measured in one research procedure at the time of the procedure. These will be compared to measurements of number and location made in the clinical surgery procedure and to measurements from clinical imaging.

SECONDARY OUTCOMES:
Size of stones determined with research ultrasound vs. clinically. The outcome measured will be the accuracy new ultrasound images versus existing clinical data. | Research data are collected on Day 1 (the day of the research imaging procedure). Clinical data are also available on Day 1. Clinical data will be downloaded by Day 7, and comparison will be made by Day 14.
  The size of stones will be measured in one research procedure at the time of the procedure. These will be compared to measurements of number and location made in the clinical surgery procedure and to measurements from clinical imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bailey, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Department of Urology, Seattle, Washington, United States

REFERENCES:
- [Result] May PC, Haider Y, Dunmire B, Cunitz BW, Thiel J, Liu Z, Bruce M, Bailey MR, Sorensen MD, Harper JD. Stone-Mode Ultrasound for Determining Renal Stone Size. J Endourol. 2016 Sep;30(9):958-62. doi: 10.1089/end.2016.0341. PMID 27393000
- [Result] Cunitz BW, Harper JD, Sorensen MD, Haider YA, Thiel J, May PC, Liu Z, Bailey MR, Dunmire B, Bruce M. Quantification of Renal Stone Contrast with Ultrasound in Human Subjects. J Endourol. 2017 Nov;31(11):1123-1130. doi: 10.1089/end.2017.0404. Epub 2017 Sep 28. PMID 28847171

DOCUMENTS (1):
  • Study Protocol (2025-07-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT02214836/Prot_000.pdf